CLINICAL TRIAL: NCT03287791
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Vehicle-Controlled Study to Evaluate Safety and Clinical Equivalence of a Generic Azelaic Acid Foam, 15% and the Reference Listed Finacea® (Azelaic Acid) Foam,15% in Patients With Moderate Facial Rosacea
Brief Title: A Study to Evaluate Safety and Equivalence of Generic Azelaic Acid Foam and Finacea® Foam in Participants With Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTA/AZEL/2015
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — azelaic acid; Sunscreening Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Generic Azelaic Acid Foam (Experimental): A thin layer of generic azelaic acid, 15% topical foam was to be gently massaged into the entire facial area twice daily, once in the morning and once in the evening, for 12 weeks. Contact with the mouth, eyes, and other mucous membranes was to be avoided. Hands were to be washed following application of study drug. Participants were instructed not to bathe, shower, wash, or swim for at least 4 hours after application of study drug. Participants were provided with mild cleanser, a towel, sunscreen, and moisturizing lotion to be used on treated areas while participating in the study.
  Interventions: Drug: Generic Azelaic Acid Foam; Other: Cleanser; Other: Sunscreen; Other: Towel; Other: Moisturizing Lotion
- Finacea® (Azelaic Acid) Foam (Active Comparator): A thin layer of Finacea (azelaic acid), 15% topical foam was to be gently massaged into the entire facial area twice daily, once in the morning and once in the evening, for 12 weeks. Contact with the mouth, eyes, and other mucous membranes was to be avoided. Hands were to be washed following application of study drug. Participants were instructed not to bathe, shower, wash, or swim for at least 4 hours after application of study drug. Participants were provided with mild cleanser, a towel, sunscreen, and moisturizing lotion to be used on treated areas while participating in the study.
  Interventions: Drug: Finacea® (Azelaic Acid) Foam; Other: Cleanser; Other: Sunscreen; Other: Towel; Other: Moisturizing Lotion
- Vehicle Foam (Placebo Comparator): A thin layer of the vehicle topical foam was to be gently massaged into the entire facial area twice daily, once in the morning and once in the evening, for 12 weeks. Contact with the mouth, eyes, and other mucous membranes was to be avoided. Hands were to be washed following application of study drug. Participants were instructed not to bathe, shower, wash, or swim for at least 4 hours after application of study drug. Participants were provided with mild cleanser, a towel, sunscreen, and moisturizing lotion to be used on treated areas while participating in the study.
  Interventions: Drug: Vehicle Foam; Other: Cleanser; Other: Sunscreen; Other: Towel; Other: Moisturizing Lotion

INTERVENTIONS:
Drug: Generic Azelaic Acid Foam — Topical foam, generic formulation of the brand product.
  Arms: Generic Azelaic Acid Foam
Drug: Finacea® (Azelaic Acid) Foam — Topical foam, brand product.
  Arms: Finacea® (Azelaic Acid) Foam
Drug: Vehicle Foam — Topical foam, placebo. Has no active ingredient.
  Arms: Vehicle Foam
Other: Cleanser — A mild cleanser provided to participants, so they can wash their face prior to applying the study drug.
Other: Sunscreen — Sunscreen provided to participants, so they can apply it to their face when outdoors.
Other: Towel — A soft towel provided to participants, so they can pat their face dry after washing and prior to applying the study drug.
Other: Moisturizing Lotion — Moisturizing lotion provided to participants, so they can apply it to their face, as needed.

SUMMARY:
The objectives of this study were to compare the safety and efficacy profiles of a generic Azelaic Acid Foam, 15% to the reference listed Finacea® (azelaic acid) Foam, 15% and to demonstrate therapeutic equivalence and safety of the two active foams in the treatment of moderate facial rosacea, and to demonstrate superiority of the Reference and Test products over the Vehicle.

DETAILED DESCRIPTION:
Topical azelaic acid is used to treat inflammatory papules and pustules of mild to moderate rosacea. Other topical therapies and oral antibiotics are also used to treat rosacea symptoms. Finacea® (azelaic acid) Foam, 15% contains azelaic acid, a naturally occurring saturated dicarboxylic acid that has proven anti-inflammatory effects, as well as anti-keratinizing and antimicrobial actions.

ELIGIBILITY:
Inclusion Criteria:

* Participants had to be willing and able to provide written informed consent for the study
* Healthy males or non-pregnant females ≥18 years-of-age with a clinical diagnosis of moderate facial rosacea
* Participants had to have at least 8 and not more than 50 inflammatory facial lesions (that is, papules/pustules) and ≤2 nodules on the face. For the purposes of study treatment and evaluation, these lesions were limited to the facial treatment area including those present on the nose. Lesions involving the eyes and scalp were excluded from the count.
* Participants had to have persistent erythema on the face with moderate (3) score
* Participants had to have a mild (1) to moderate (2) score for telangiectasia on the face
* Participants had to have a definite clinical diagnosis of moderate facial rosacea (severity score 3)
* Participants had to be willing to minimize external factors that might trigger rosacea flare-ups (for example, spicy foods, thermally hot foods and drinks, hot environments, prolonged sun exposure, strong winds, and alcoholic beverages) during the course of the study
* Participants had to be in general good health and free from any clinically significant disease other than rosacea on the face, that could have interfered with the study evaluations
* Participants had to be willing and able to understand and comply with the requirements of the study, apply the medication as instructed, return for the required treatment period visits, comply with therapy prohibitions, and able to complete the study
* Male participants and female participants of childbearing potential had to use accepted methods of birth control or had to agree to practice abstinence, from study start to 30 days after the last administration of study drug. All female participants were considered to be of childbearing potential unless they had been surgically sterilized (hysterectomy, bilateral oophorectomy, or tubal ligation) or had been postmenopausal for at least a year. Any of the following methods of birth control were acceptable: oral contraceptives, contraceptive patches/implants (for example, Norplant®), vaginal ring (NuvaRing®), Depo-Provera® (Medroxy progesterone acetate), double barrier methods (for example, condom and spermicide), or intrauterine device
* Female participants of child bearing potential had to have a negative urine pregnancy test at baseline
* Participants who used make-up had to have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and had to agree to use the same make-up, brand/type, or frequency of use, throughout the study

Exclusion Criteria:

* Pregnant or lactating or planning to become pregnant during the study period
* Presence of any skin condition on the face that could have interfered with the diagnosis or assessment of rosacea
* Excessive facial hair (for example, beards, sideburns, moustaches) that would interfere could have interfered with diagnosis or assessment of rosacea
* History of hypersensitivity or allergy to azelaic acid, propylene glycol, or any other component of the formulation
* The use within 6 months prior to baseline of oral retinoids (for example, Accutane®) or therapeutic Vitamin A supplements of greater than 10,000 units/day (multivitamins were allowed)
* The use of estrogens or oral contraceptives for less than 3 months prior to baseline
* The use within 1 month prior to baseline of the following:

  * topical retinoids to the face
  * systemic antibiotics known to have an impact on the severity of facial rosacea (for example, containing tetracycline and its derivatives, erythromycin and its derivatives, sulfamethoxazole, or trimethoprim)
  * systemic corticosteroids
* Use within two weeks prior to baseline of the following:

  * topical corticosteroids
  * topical antibiotics
  * topical medications for rosacea (for example, metronidazole, azelaic acid)
* Antipruritics, including antihistamines, within 24 hours of any study visit
* Participants with moderate or severe rhinophyma, dense telangiectasia (score 3, severe), or plaque-like facial edema
* Participants with a severe irritation grade for erythema, dryness, scaling, pruritus, stinging/burning, and edema
* Ocular rosacea (for example, conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical or systemic antibiotics
* A participant who had used a sauna during the 2 weeks prior to study entry and during the study
* Participants who had performed wax epilation of the face within 14 days prior to baseline
* A participant who had a history of being unresponsive to topical azelaic acid therapy
* A participant who had any clinically significant condition or situation, other than the condition being studied that, in the opinion of the Investigator, could have interfered with the study evaluations or optimal participation in the study
* A participant who had used any topical azelaic acid therapy within 30 days of baseline visit
* Participants who had participated in an investigational drug study (for example, participants had been treated with an investigational drug) within 30 days prior to baseline were excluded from study participation. Participants who were participating in non-treatment studies such as observational studies or registry studies could be considered for inclusion
* Participants who had been previously randomized in this study
* Participants who had laser therapy (for telangiectasia or other conditions) and phototherapy to the facial area within 180 days prior to study entry
* Participants who had cosmetic procedures (for example, facials), which could affect the efficacy and safety profile of the investigational product within 14 days prior to study entry
* Employees or staff of the research site were excluded from participation in the study
* No more than 1 participant from the same household was allowed to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 924 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Teva Pharmaceuticals USA
Locations (26):
- United States (26):
  - Investigative Site 2, Encino, California
  - Investigative Site 10, La Mesa, California
  - Investigative Site 19, Brandon, Florida
  - Investigative Site 1, Hialeah, Florida
  - Investigative Site 9, Hialeah, Florida
  - Investigative Site 23, Lauderdale Lakes, Florida
  - Investigative Site 11, Miami, Florida
  - Investigative Site 15, Miami, Florida
  - Investigative Site 20, Miami, Florida
  - Investigative Site 12, Miramar, Florida
  - Investigative Site 25, Ocala, Florida
  - Investigative Site 22, Pembroke Pines, Florida
  - Investigative Site 18, Tampa, Florida
  - Investigative Site 16, Savannah, Georgia
  - Investigative Site 14, Plainfield, Indiana
  - Investigative Site 13, Wichita, Kansas
  - Investigative Site 6, New Orleans, Louisiana
  - Investigative Site 17, Omaha, Nebraska
  - Investigative Site 8, High Point, North Carolina
  - Investigative Site 3, Cincinnati, Ohio
  - Investigative Site 21, Philadelphia, Pennsylvania
  - Investigative Site 4, Dallas, Texas
  - Investigative Site 26, El Paso, Texas
  - Investigative Site 7, New Braunfels, Texas
  - Investigative Site 5, Norfolk, Virginia
  - Investigative Site 24, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The populations for this study included the Safety Population, the modified Intent-to-Treat (mITT) population, and the Per-Protocol (PP) Population.
Pre-assignment Details: If participant failed to return diary card and had no evidence of study drug use, then •participant was included in Safety population if there was some participant safety or efficacy data after Baseline •participant considered lost to follow up and excluded from Safety Population if there was no participant safety or efficacy data after Baseline
Groups:
- Generic Azelaic Acid Foam: A thin layer of generic azelaic acid, 15% topical foam was to be gently massaged into the entire facial area twice daily, once in the morning and once in the evening, for 12 weeks (wks). Contact with the mouth, eyes, and other mucous membranes was to be avoided. Hands were to be washed following application of study drug. Participants were instructed not to bathe, shower, wash, or swim for at least 4 hours after application of study drug. Participants were provided with mild cleanser, a towel, sunscreen, and moisturizing lotion to be used on treated areas while participating in the study.
- Finacea (Azelaic Acid) Foam: A thin layer of Finacea (azelaic acid), 15% topical foam was to be gently massaged into the entire facial area twice daily, once in the morning and once in the evening, for 12 weeks. Contact with the mouth, eyes, and other mucous membranes was to be avoided. Hands were to be washed following application of study drug. Participants were instructed not to bathe, shower, wash, or swim for at least 4 hours after application of study drug. Participants were provided with mild cleanser, a towel, sunscreen, and moisturizing lotion to be used on treated areas while participating in the study.
Period: Overall Study
Arm/Group | Generic Azelaic Acid Foam | Finacea (Azelaic Acid) Foam | Vehicle Foam
Started | 312 | 312 | 300
Safety Population (Randomized participants with evidence in diary card of using ≥1 dose of study drug.) | 306 | 297 | 291
mITT Population (Safety Population, met inclusion/exclusion criteria, have ≥1 post-baseline efficacy data) | 291 | 291 | 283
PP Population (mITT, >75-125% doses and >6 consecutive doses, or discontinued for lack of treatment-completed ≥8wks) | 262 | 259 | 245
Completed | 280 | 276 | 264
Not Completed | 32 | 36 | 36
Not completed — Insufficient Therapeutic Response | 0 | 0 | 1
Not completed — Adverse Event | 0 | 4 | 3
Not completed — Withdrawal by Subject | 12 | 12 | 17
Not completed — Missed more than 6 consecutive doses | 3 | 2 | 2
Not completed — Lost to Follow-up | 8 | 14 | 11
Not completed — Protocol Violation | 7 | 2 | 1
Not completed — Participant was enrolled at 2 sites | 1 | 0 | 1
Not completed — Too much time between 2 visits | 0 | 1 | 0
Not completed — Non-compliance | 0 | 1 | 0
Not completed — Did not meet inclusion criteria | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants with evidence in diary card of using ≥1 dose of study drug (Safety Population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Azelaic Acid Foam | Finacea (Azelaic Acid) Foam | Vehicle Foam | Total
Number analyzed (Participants) | 306 | 297 | 291 | 894
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (14.20) | 52.3 (15.14) | 51.0 (15.09) | 51.6 (14.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 220 | 204 | 636
  Male | 94 | 77 | 87 | 258
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 185 | 177 | 180 | 542
  Not Hispanic or Latino | 121 | 120 | 111 | 352
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 3 | 11
  White | 302 | 292 | 288 | 882
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Inflammatory Lesion Count [Mean (Standard Deviation); unit: inflammatory lesions] — All facial papules and pustules were considered inflammatory lesions. Papule defined as inflammatory lesion; small (≤5 millimeters [mm] in diameter), solid palpable lesion, usually with inflamed elevation of the skin that does not contain pus. Pustule defined as inflammatory lesion; small (≤5 mm in diameter), inflamed skin swelling that is filled with pus.
  inflammatory lesions | 17.1 (8.85) | 16.7 (7.88) | 17.7 (8.88) | 17.1 (8.55)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Inflammatory Lesions (Papules and Pustules) Counts at Week 12
Description: All facial papules, pustules, and nodules, located above the jaw line and extending to the hairline, were counted. When counting facial lesions, lesions present on the nose were included. The total count for each lesion type was recorded and the total number of inflammatory lesions (papules and pustules) were calculated. A papule with a pustule on its apex was counted as a pustule. Counts of nodules and cysts were reported separately and not included in the inflammatory counts. Papule defined as inflammatory lesion; small (≤5 mm in diameter), solid palpable lesion, usually with inflamed elevation of the skin that does not contain pus. Pustule defined as inflammatory lesion; small (≤5 mm in diameter), inflamed skin swelling that is filled with pus. Cyst and nodule defined as palpable solid or soft lesion >5 mm in diameter.
Time Frame: Baseline, 12 weeks
Population: Participants in the PP Population. If participant discontinued between 8 and 12 weeks of treatment due to lack of treatment, last observation carried forward (LOCF) was used to impute the number of lesions. If participant was missing Week 12 assessment for any other reason, participant was excluded.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Generic Azelaic Acid Foam | Finacea (Azelaic Acid) Foam | Vehicle Foam
Number analyzed (Participants) | 262 | 259 | 245
percent change | -64.28 (25.050) | -65.15 (26.419) | -57.84 (30.626)
Statistical Analysis 1: Comparison: Generic Azelaic Acid Foam vs Vehicle Foam; Analyses was performed using an Analysis of Variance (ANOVA) model with percent change from baseline to Week 12 in the lesion count as outcome and treatment, center and treatment-by-center interaction as factors; Test type: Superiority; p < .0001, ANOVA; Mean Difference (Final Values) = -11.27, 95% CI 2-sided [-16.80 to -5.73]
Statistical Analysis 2: Comparison: Finacea (Azelaic Acid) Foam vs Vehicle Foam; Analyses was performed using an ANOVA model with percent change from baseline to Week 12 in the lesion count as outcome and treatment, center and treatment-by-center interaction as factors; Test type: Superiority; p = 0.0007, ANOVA; Median Difference (Final Values) = -9.71, 95% CI 2-sided [-15.28 to -4.14]

2. Secondary Outcome: Percentage of Participants With Treatment Success Based on IGE Score
Description: Treatment success defined as an Investigator's Global Evaluation (IGE) score at Week 12 of 0 (clear) or 1 (almost clear). Any other outcome was considered a failure. Participants who were discontinued prematurely from the study due to lack of treatment effect after at least 8 weeks of compliant treatment were considered as treatment failures. The IGE score was based on a 5-point scale ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe).
Time Frame: Baseline and 12 Weeks
Population: Participants in the PP Population. Participants who did not have a valid Week 12 assessment for any other reason were excluded from the PP analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Generic Azelaic Acid Foam | Finacea (Azelaic Acid) Foam | Vehicle Foam
Number analyzed (Participants) | 262 | 259 | 245
percentage of participants | 39.7 | 48.3 | 33.5

ADVERSE EVENTS:
Time Frame: Baseline up to Day 84
Description: Adverse events were collected from participants who were randomized and had evidence in diary card of using ≥1 dose of study drug (Safety Population).
Arm/Group | Generic Azelaic Acid Foam | Finacea (Azelaic Acid) Foam | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/306 | 0/297 | 0/291
Serious Adverse Events (participants affected / at risk) | 0/306 | 2/297 | 1/291
Other Adverse Events (participants affected / at risk) | 129/306 | 128/297 | 125/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Generic Azelaic Acid Foam (N=306) | Finacea (Azelaic Acid) Foam (N=297) | Vehicle Foam (N=291)
Prostate cancer (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Azelaic Acid Foam (N=306) | Finacea (Azelaic Acid) Foam (N=297) | Vehicle Foam (N=291)
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Application site acne (General disorders) | 1 | 0 | 0
Application site dryness (General disorders) | 45 | 29 | 52
Application site erythema (General disorders) | 30 | 28 | 34
Application site exfoliation (General disorders) | 1 | 0 | 1
Application site inflammation (General disorders) | 0 | 0 | 1
Application site irritation (General disorders) | 0 | 1 | 1
Application site oedema (General disorders) | 3 | 4 | 5
Application site pain (General disorders) | 47 | 41 | 28
Application site pruritus (General disorders) | 51 | 43 | 28
Application site reaction (General disorders) | 22 | 19 | 20
Application site swelling (General disorders) | 2 | 6 | 8
Application site vesicles (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Application site folliculitis (Infections and infestations) | 0 | 1 | 0
Application site pustules (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 6 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 4 | 3
Oral herpes (Infections and infestations) | 1 | 0 | 0
Pertussis (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Biopsy skin (Investigations) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 15 | 9 | 12
Migraine (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of Multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT03287791/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03287791/SAP_001.pdf